CLINICAL TRIAL: NCT01259154
Title: Combined Bipolar Radiofrequency Surgery of the Tongue Base and Uvulopalatopharyngoplasty for Obstructive Sleep Apnea
Brief Title: Combined RF Surgery of the Tongue Base and Uvulopalatopharyngoplasty (UPPP) for Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Other Study IDs: CU123
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-12

CONDITIONS: Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- RFITT+UPPP
- UPPP

SUMMARY:
Introduction: The aim of the study was to investigate the effectiveness of combined bipolar radiofrequency surgery of the tongue base (RFBT) and uvulopalatopharyngoplasty (UPPP) in a single session for obstructive sleep apnea (OSA) and to determine whether this combination is safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria: obstructive sleep apnea not treated by CPAP

Exclusion Criteria: a history of previous surgery for OSA and only one level of airway obstruction

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with obstructive sleep apnea not treated by CPAP
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty Hospital Motol, Prague, Czechia